CLINICAL TRIAL: NCT01936285
Title: Study of Anti-inflammatory Treatment With Colchicine in the Acute Phase of ST-elevation Myocardial Infarction to Reduce Infarct Size
Brief Title: Colchicine in ST-elevation Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: G.Gennimatas General Hospital (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Director, Cardiac Catheterization Department, G.Gennimatas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COL.ACS
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Colchicine; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): Patients taking placebo
  Interventions: Drug: Placebo
- Colchicine (Experimental): Active treatment group
  Interventions: Drug: Colchicine 2 mg loading dose; 0.5 mg bid for 5 days

INTERVENTIONS:
Drug: Colchicine 2 mg loading dose; 0.5 mg bid for 5 days
  Arms: Colchicine
Drug: Placebo
  Arms: Control group

SUMMARY:
* There is evidence that inflammatory processes may play detrimental role during the acute phase of myocardial infarction
* The hypothesis of this study is that colchicine, by its anti-inflammatory action, may lead to reduction in infarct size, when administered during the acute phase of myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

The study will enroll patients 18 years old or older who present to the hospital within twelve (12) hours of the onset of chest pain and who had ST segment elevation >1 mm in two contiguous limb leads or ST segment elevation >2 mm in two consecutive precordial leads or new onset of left bundle branch block (LBBB) in a twelve lead electrocardiogram and for whom the decision was made to be taken to the cath lab to perform angioplasty of the coronary vessels.

Excluded patients:

* > 80 years old
* with active inflammatory diseases, infectious diseases or known malignancy
* under treatment with corticosteroids, anti-inflammatory agents or disease modifying agents
* with known hypersensitivity-allergy to colchicine
* under chronic treatment with colchicine
* with severe renal failure (eGFR < 30 ml/min/1.73 m2)
* with hepatic failure (Child - Pugh class B or C)
* presenting with cardiac arrest
* presenting with ventricular fibrillation
* presenting with cardiogenic shock
* with stent thrombosis
* with angina within 48 hours before infarction
* with previous myocardial infarction
* with occlusion of the left main or left circumflex coronary artery or with evidence of coronary collaterals to the region at risk on initial coronary angiography (at the time of admission)
* with metallic implants (ferromagnetic material)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Infarct size on MRI | 5 days post-MI
  MRI with LGE will be performed in a subset of study participants
AUC CK-MB concentration | 0-3 days post-MI
  Area under the curve of creatine kinase-MB fraction concentrations from presentation to 72h will be assessed in all recruits

SECONDARY OUTCOMES:
Myocardial damage marker levels | Days 1-3 post-MI
  Maximal concentrations of hs-TnT and CK-MB

CONTACTS AND LOCATIONS:
Locations (1):
- Athens General Hospital "G. Gennimatas", Athens, Greece

REFERENCES:
- [Derived] Deftereos S, Giannopoulos G, Angelidis C, Alexopoulos N, Filippatos G, Papoutsidakis N, Sianos G, Goudevenos J, Alexopoulos D, Pyrgakis V, Cleman MW, Manolis AS, Tousoulis D, Lekakis J. Anti-Inflammatory Treatment With Colchicine in Acute Myocardial Infarction: A Pilot Study. Circulation. 2015 Oct 13;132(15):1395-403. doi: 10.1161/CIRCULATIONAHA.115.017611. Epub 2015 Aug 11. PMID 26265659